CLINICAL TRIAL: NCT04770155
Title: Vascular Dysfunction in Black Individuals: Roles of Nitric Oxide and Endothelin-1
Acronym: UMMC_Pilot
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Despite significant effort, we were unable to obtain the supply of drugs and supplements needed for the various arms of this Clinical Trial.
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Thales Coelho Barbosa, Instructor, University of Mississippi Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2P20GM104357-08 (NIH)
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Vascular Function; Racial Disparity
Keywords: Black; African American; White; Caucasian American; Hyperemia; Blood Flow; Conductance
MeSH Terms: conditions — Hyperemia | interventions — Citrulline; Sildenafil Citrate; Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Beetroot juice (Aim 1a) (Active Comparator): Upon arriving at the laboratory, participants will ingest 140 ml of beetroot juice containing a high (~12.8 mmol) concentration of nitrates (James White Drinks, Suffolk, UK).
  Interventions: Dietary Supplement: Dietary Nitrates 400 mg
- Placebo (Aim 1a) (Placebo Comparator): Upon arriving at the laboratory, participants will ingest 140 ml of beetroot juice containing a low concentration (~0.0055 mmol) of nitrates (James White Drinks, Suffolk, UK).
  Interventions: Dietary Supplement: Dietary Nitrates 400 mg
- L-citrulline (Aim 1b) (Active Comparator): Participants will receive pills containing 3 g of L-citrulline (Superior Labs, Park City, UT) to take twice daily for 7 days before the study visit.
  Interventions: Dietary Supplement: L-citrulline 3 g
- Placebo (Aim 1b) (Placebo Comparator): Participants will receive pills containing a placebo to take twice daily for 7 days before the study visit.
  Interventions: Dietary Supplement: L-citrulline 3 g
- Sildenafil (Aim 1c) (Active Comparator): Upon arriving at the laboratory, participants will ingest a liquid mixture containing Sildenafil (100 mg), an inhibitor of phosphodiesterase 5.
  Interventions: Drug: Sildenafil 100 mg
- Placebo (Aim 1c) (Placebo Comparator): Upon arriving at the laboratory, participants will ingest a liquid mixture containing a placebo.
  Interventions: Drug: Sildenafil 100 mg
- Bosentan (Aim 2) (Active Comparator): Upon arriving at the laboratory, participants will ingest a liquid mixture containing Bosentan (125 mg), a non-selective blocker of endothelin-1 receptors ETA and ETB.
  Interventions: Drug: Bosentan 125 mg
- Placebo (Aim 2) (Placebo Comparator): Upon arriving at the laboratory, participants will ingest a liquid mixture containing a placebo.
  Interventions: Drug: Bosentan 125 mg

INTERVENTIONS:
Dietary Supplement: Dietary Nitrates 400 mg — The nitrates in the beetroot juice will be absorbed and reduced in the plasma to nitrite and nitric oxide, increasing endothelium-independent nitric oxide bioavailability.
  Other Names: Beet It Sport Nitrate 400
  Arms: Beetroot juice (Aim 1a); Placebo (Aim 1a)
Dietary Supplement: L-citrulline 3 g — Ingested L-citrulline becomes available in large quantities in the plasma for enzymatic conversion into L-arginine. The activity of the endothelial nitric oxide synthase converts L-arginine into nitric oxide, increasing endothelium-dependent nitric oxide bioavailability.
  Arms: L-citrulline (Aim 1b); Placebo (Aim 1b)
Drug: Sildenafil 100 mg — Sildenafil inhibits phosphodiesterase 5, an enzyme that degrades cyclic guanosine monophosphate in the vascular smooth muscle cells inactivating the nitric oxide-mediated signal; thus, Sildenafil will prolong the availability of cyclic guanosine monophosphate, enhancing the nitric oxide-mediated intracellular cascade.
  Other Names: Viagra, Revatio
  Arms: Placebo (Aim 1c); Sildenafil (Aim 1c)
Drug: Bosentan 125 mg — Bosentan blocks endothelin-1 receptors ETA and ETB, leading to a reduction in vasoconstrictor tone and a greater magnitude of vasodilator responses.
  Other Names: Tracleer
  Arms: Bosentan (Aim 2); Placebo (Aim 2)

SUMMARY:
The research aims of this proposal are:

* Specific Aim 1: To test whether an increase in nitric oxide signaling can increase vasodilator responses in young Black individuals.
* Specific Aim 2: To test whether a decrease in endothelin-1 signaling can increase vasodilator responses in young Black individuals.

DETAILED DESCRIPTION:
Studies will be conducted in the Clinical Research and Trials Unit at the University of Mississippi Medical Center. All study visits will follow the same procedures, except for the drug or supplement being administered.

For Aim 1, double-blind, randomized, placebo-controlled crossover designs will examine the effects of increasing nitric oxide and cyclic guanosine monophosphate bioavailability on vascular function of young Black and White individuals. Three sets of two visits will be performed:

* Aim 1a: At the beginning of each visit, participants will ingest either a nitrate-rich beetroot juice or a nitrate-depleted beetroot juice (serving as placebo) in their liquid commercial form, which has a distinct color and flavor. The nitrates will be absorbed and reduced in the plasma to nitrite and nitric oxide, increasing endothelium-independent nitric oxide bioavailability.
* Aim 1b: Participants will receive a 7-day supplement of L-citrulline or placebo before each study visit, with a washout period of 7 days between visits. The activity of the endothelial nitric oxide synthase converts L-arginine into nitric oxide and L-citrulline, which is normally recycled back into L-arginine. Unlike L-arginine, oral ingestion of L-citrulline is not catabolized in the gut, nor is it extracted from systemic circulation through hepatic first-pass metabolism. Thus, ingested L-citrulline becomes available in large quantities in the plasma for enzymatic conversion into L-arginine, increasing endothelium-dependent nitric oxide bioavailability.
* Aim 1c: At the beginning of each visit, participants will ingest a liquid mixture prepared by Investigational Drug Services at the University of Mississippi Medical Center containing Sildenafil or placebo. Sildenafil inhibits phosphodiesterase 5, an enzyme that degrades cyclic guanosine monophosphate in the vascular smooth muscle cells inactivating the nitric oxide-mediated signal; thus, Sildenafil will prolong the availability of cyclic guanosine monophosphate, enhancing the nitric oxide-mediated intracellular cascade.

For Aim 2, a double-blind, randomized, placebo-controlled crossover design will examine the role of endothelin-1 on the vascular function of young Black and White individuals. Two visits will be performed, with a minimum of 7 days between them.

• Aim 2: At the beginning of each visit, participants will ingest a liquid mixture prepared by Investigational Drug Services at the University of Mississippi Medical Center containing Bosentan or placebo. Bosentan blocks ETA and ETB receptors, leading to a reduction in vasoconstrictor tone and a greater magnitude of vasodilator responses.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification of their race and the race of their biological parents as being only Black (i.e., African American) or only White (i.e., Caucasian American)
* Born and raised in the United States

Exclusion Criteria:

* Mixed races
* Any chronic or ongoing disease
* Prescribed pharmacological treatment
* Smoking or tobacco use
* Obesity (body mass index > 30 kg / m2)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thales C Barbosa, Ph.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
Doppler ultrasound videos, analog-digital recordings, participants' characteristics, and randomization codes will be available in an unidentified format.
Supporting Information: Study Protocol
Time Frame: On Jan 1st, 2025 for one year.
Access Criteria: By request.

REFERENCES:
- [Background] Barbosa TC, Young BE, Stephens BY, Nandadeva D, Kaur J, Keller DM, Fadel PJ. Functional sympatholysis is preserved in healthy young Black men during rhythmic handgrip exercise. Am J Physiol Regul Integr Comp Physiol. 2020 Sep 1;319(3):R323-R328. doi: 10.1152/ajpregu.00105.2020. Epub 2020 Aug 12. PMID 32783690
- [Background] Barbosa TC, Kaur J, Stephens BY, Akins JD, Keller DM, Brothers RM, Fadel PJ. Attenuated forearm vascular conductance responses to rhythmic handgrip in young African-American compared with Caucasian-American men. Am J Physiol Heart Circ Physiol. 2018 Nov 1;315(5):H1316-H1321. doi: 10.1152/ajpheart.00387.2018. Epub 2018 Aug 17. PMID 30118345
- [Background] Kaur J, Barbosa TC, Nandadeva D, Young BE, Stephens BY, Brothers RM, Fadel PJ. Attenuated Rapid-Onset Vasodilation to Forearm Muscle Contraction in Black Men. Med Sci Sports Exerc. 2021 Mar 1;53(3):590-596. doi: 10.1249/MSS.0000000000002511. PMID 32910095
- [Background] Young BE, Kaur J, Vranish JR, Stephens BY, Barbosa TC, Cloud JN, Wang J, Keller DM, Fadel PJ. Augmented resting beat-to-beat blood pressure variability in young, healthy, non-Hispanic black men. Exp Physiol. 2020 Jul;105(7):1102-1110. doi: 10.1113/EP088535. Epub 2020 May 27. PMID 32362031
- [Background] Vranish JR, Holwerda SW, Young BE, Credeur DP, Patik JC, Barbosa TC, Keller DM, Fadel PJ. Exaggerated Vasoconstriction to Spontaneous Bursts of Muscle Sympathetic Nerve Activity in Healthy Young Black Men. Hypertension. 2018 Jan;71(1):192-198. doi: 10.1161/HYPERTENSIONAHA.117.10229. Epub 2017 Dec 4. PMID 29203629

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Beetroot Juice, Then Placebo (Aim 1a): Upon arriving at the laboratory, participants will ingest 140 ml of beetroot juice containing a high (~12.8 mmol) concentration of nitrates (James White Drinks, Suffolk, UK), or 140 ml of beetroot juice containing a low concentration (~0.0055 mmol) of nitrates (James White Drinks, Suffolk, UK).
  Dietary Nitrates 400 mg: The nitrates in the beetroot juice will be absorbed and reduced in the plasma to nitrite and nitric oxide, increasing endothelium-independent nitric oxide bioavailability.
- Experimental: Placebo, Then Beetroot Juice (Aim 1a): Upon arriving at the laboratory, participants will ingest 140 ml of beetroot juice containing a low concentration (~0.0055 mmol) of nitrates (James White Drinks, Suffolk, UK), or 140 ml of beetroot juice containing a high (~12.8 mmol) concentration of nitrates (James White Drinks, Suffolk, UK).
  Dietary Nitrates 400 mg: The nitrates in the beetroot juice will be absorbed and reduced in the plasma to nitrite and nitric oxide, increasing endothelium-independent nitric oxide bioavailability.
- Experimental: L-citrulline, Then Placebo (Aim 1b): Participants will receive pills containing 3 g of L-citrulline (Superior Labs, Park City, UT) to take twice daily for 7 days before the study visit, or pills containing a placebo to take twice daily for 7 days before the study visit.
  L-citrulline 3 g: Ingested L-citrulline becomes available in large quantities in the plasma for enzymatic conversion into L-arginine. The activity of the endothelial nitric oxide synthase converts L-arginine into nitric oxide, increasing endothelium-dependent nitric oxide bioavailability.
- Experimental: Placebo, Then L-citrulline (Aim 1b): Participants will receive pills containing a placebo to take twice daily for 7 days before the study visit, or pills containing 3 g of L-citrulline (Superior Labs, Park City, UT) to take twice daily for 7 days before the study visit.
  L-citrulline 3 g: Ingested L-citrulline becomes available in large quantities in the plasma for enzymatic conversion into L-arginine. The activity of the endothelial nitric oxide synthase converts L-arginine into nitric oxide, increasing endothelium-dependent nitric oxide bioavailability.
- Experimental: Sildenafil, Then Placebo (Aim 1c): Upon arriving at the laboratory, participants will ingest a liquid mixture containing Sildenafil (100 mg), an inhibitor of phosphodiesterase 5, or a liquid mixture containing a placebo.
  Sildenafil 100 mg: Sildenafil inhibits phosphodiesterase 5, an enzyme that degrades cyclic guanosine monophosphate in the vascular smooth muscle cells inactivating the nitric oxide-mediated signal; thus, Sildenafil will prolong the availability of cyclic guanosine monophosphate, enhancing the nitric oxide-mediated intracellular cascade.
- Experimental: Placebo, Then Sildenafil (Aim 1c): Upon arriving at the laboratory, participants will ingest a liquid mixture containing a placebo, or a liquid mixture containing Sildenafil (100 mg), an inhibitor of phosphodiesterase 5.
  Sildenafil 100 mg: Sildenafil inhibits phosphodiesterase 5, an enzyme that degrades cyclic guanosine monophosphate in the vascular smooth muscle cells inactivating the nitric oxide-mediated signal; thus, Sildenafil will prolong the availability of cyclic guanosine monophosphate, enhancing the nitric oxide-mediated intracellular cascade.
- Experimental: Bosentan, Then Placebo (Aim 2): Upon arriving at the laboratory, participants will ingest a liquid mixture containing Bosentan (125 mg), a non-selective blocker of endothelin-1 receptors ETA and ETB, or a liquid mixture containing a placebo.
  Bosentan 125 mg: Bosentan blocks endothelin-1 receptors ETA and ETB, leading to a reduction in vasoconstrictor tone and a greater magnitude of vasodilator responses.
- Experimental: Placebo, Then Bosentan (Aim 2): Upon arriving at the laboratory, participants will ingest a liquid mixture containing a placebo, or a liquid mixture containing Bosentan (125 mg), a non-selective blocker of endothelin-1 receptors ETA and ETB.
  Bosentan 125 mg: Bosentan blocks endothelin-1 receptors ETA and ETB, leading to a reduction in vasoconstrictor tone and a greater magnitude of vasodilator responses.
Period: Overall Study
Arm/Group | Experimental: Beetroot Juice, Then Placebo (Aim 1a) | Experimental: Placebo, Then Beetroot Juice (Aim 1a) | Experimental: L-citrulline, Then Placebo (Aim 1b) | Experimental: Placebo, Then L-citrulline (Aim 1b) | Experimental: Sildenafil, Then Placebo (Aim 1c) | Experimental: Placebo, Then Sildenafil (Aim 1c) | Experimental: Bosentan, Then Placebo (Aim 2) | Experimental: Placebo, Then Bosentan (Aim 2)
Started (The only data collected were baseline measurements and no participants were ever given either intervention; the investigator was never able to obtain the treatments to use for the planned intervention arm of the study, resulting in its termination.) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed (The only data collected were baseline measurements and no participants were ever given either intervention; the investigator was never able to obtain the treatments to use for the planned intervention arm of the study, resulting in its termination.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not completed — Baseline measurements only. Investigator did not obtain treatments for the planned interventions. | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The only data collected were baseline measurements and no participants were ever given either intervention; the investigator was never able to obtain the treatments to use for the planned intervention arm of the study, resulting in its termination. Upon resigning of his Instructor position at UMMC, the investigator backed up the baseline data files on an external hard drive. Unfortunately, some issue with the external hard drive corrupted the files, making them no longer accessible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Beetroot Juice, Then Placebo (Aim 1a) | Experimental: Placebo, Then Beetroot Juice (Aim 1a) | Experimental: L-citrulline, Then Placebo (Aim 1b) | Experimental: Placebo, Then L-citrulline (Aim 1b) | Experimental: Sildenafil, Then Placebo (Aim 1c) | Experimental: Placebo, Then Sildenafil (Aim 1c) | Experimental: Bosentan, Then Placebo (Aim 2) | Experimental: Placebo, Then Bosentan (Aim 2) | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 8
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Male | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 7
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation
Description: The percent change in arterial diameter normalized to arterial shear rate during reperfusion after 5 minutes of circulatory occlusion.
Time Frame: Within 4 hours of drug/supplement administration.
Population: Flow-mediated dilation was not collected in any participant.
Arm/Group | Experimental: Beetroot Juice, Then Placebo (Aim 1a) | Experimental: Placebo, Then Beetroot Juice (Aim 1a) | Experimental: L-citrulline, Then Placebo (Aim 1b) | Experimental: Placebo, Then L-citrulline (Aim 1b) | Experimental: Sildenafil, Then Placebo (Aim 1c) | Experimental: Placebo, Then Sildenafil (Aim 1c) | Experimental: Bosentan, Then Placebo (Aim 2) | Experimental: Placebo, Then Bosentan (Aim 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Reactive Hyperemia (Cuff Release)
Description: Blood velocity area-under-the-curve from the beginning of reperfusion to return to resting values.
Time Frame: Within 4 hours of drug/supplement administration.
Population: Reactive hyperemia with cuff release was not collected in any participant.
Arm/Group | Experimental: Beetroot Juice, Then Placebo (Aim 1a) | Experimental: Placebo, Then Beetroot Juice (Aim 1a) | Experimental: L-citrulline, Then Placebo (Aim 1b) | Experimental: Placebo, Then L-citrulline (Aim 1b) | Experimental: Sildenafil, Then Placebo (Aim 1c) | Experimental: Placebo, Then Sildenafil (Aim 1c) | Experimental: Bosentan, Then Placebo (Aim 2) | Experimental: Placebo, Then Bosentan (Aim 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Muscle Hyperemia (Passive Leg Movement)
Description: Peak and the area-under-the-curve of the change in femoral artery blood flow during 1 minute of passive leg movement.
Time Frame: Within 4 hours of drug/supplement administration.
Population: Muscle hyperemia with passive leg movement was not collected in any participant.
Arm/Group | Experimental: Beetroot Juice, Then Placebo (Aim 1a) | Experimental: Placebo, Then Beetroot Juice (Aim 1a) | Experimental: L-citrulline, Then Placebo (Aim 1b) | Experimental: Placebo, Then L-citrulline (Aim 1b) | Experimental: Sildenafil, Then Placebo (Aim 1c) | Experimental: Placebo, Then Sildenafil (Aim 1c) | Experimental: Bosentan, Then Placebo (Aim 2) | Experimental: Placebo, Then Bosentan (Aim 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Muscle Hyperemia (Rhythmic Handgrip Exercise)
Description: Changes in brachial artery blood flow and conductance during single handgrip contractions at 3 intensities.
Time Frame: Baseline measurements with no drug/supplement administration before or after.
Population: The only data collected were baseline measurements and no participants were ever given either intervention; the investigator was never able to obtain the treatments to use for the planned intervention arm of the study, resulting in its termination. Upon resigning his Instructor position at UMMC, the investigator backed up the baseline data files on an external hard drive. Unfortunately, some issues with the external hard drive corrupted the files, making them no longer accessible.
Arm/Group | Experimental: Beetroot Juice, Then Placebo (Aim 1a) | Experimental: Placebo, Then Beetroot Juice (Aim 1a) | Experimental: L-citrulline, Then Placebo (Aim 1b) | Experimental: Placebo, Then L-citrulline (Aim 1b) | Experimental: Sildenafil, Then Placebo (Aim 1c) | Experimental: Placebo, Then Sildenafil (Aim 1c) | Experimental: Bosentan, Then Placebo (Aim 2) | Experimental: Placebo, Then Bosentan (Aim 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Muscle Hyperemia (Rhythmic Knee Extension Exercise)
Description: Changes in femoral artery blood flow and conductance during 3 minutes of rhythmic knee extension exercise.
Time Frame: Within 4 hours of drug/supplement administration.
Population: Muscle hyperemia with rhythmic knee extension exercise was not collected in any participant.
Arm/Group | Experimental: Beetroot Juice, Then Placebo (Aim 1a) | Experimental: Placebo, Then Beetroot Juice (Aim 1a) | Experimental: L-citrulline, Then Placebo (Aim 1b) | Experimental: Placebo, Then L-citrulline (Aim 1b) | Experimental: Sildenafil, Then Placebo (Aim 1c) | Experimental: Placebo, Then Sildenafil (Aim 1c) | Experimental: Bosentan, Then Placebo (Aim 2) | Experimental: Placebo, Then Bosentan (Aim 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed because the only data collected were baseline measurements and no participants were ever given either intervention. The investigator was never able to obtain the treatments to use for the planned intervention arm of the study, resulting in its termination.
Description: Adverse events were not assessed because the only data collected were baseline measurements and no participants were ever given either intervention. The investigator was never able to obtain the treatments to use for the planned intervention arm of the study, resulting in its termination.
Arm/Group | Beetroot Juice (Aim 1a) | Placebo (Aim 1a) | L-citrulline (Aim 1b) | Placebo (Aim 1b) | Sildenafil (Aim 1c) | Placebo (Aim 1c) | Bosentan (Aim 2) | Placebo (Aim 2)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The only data collected were baseline measurements and no participants were ever given either intervention; the investigator was never able to obtain the treatments to use for the planned intervention arm of the study, resulting in its termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04770155/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04770155/ICF_001.pdf